CLINICAL TRIAL: NCT03006939
Title: Intraoperative Fluid Balance During Cytoreductive Surgery for Ovarian Cancer
Brief Title: Fluid Balance During Surgery for Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Martin Soehle, Vice head of the department, University Hospital, Bonn
Other Study IDs: FBO
Record Dates: First submitted 2016-12-14; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Ovarian Neoplasm; Fluid Therapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are retained to determine the coagulation status as well as the albumine concentration
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cytoreductive surgery — Cytoreductive surgery in terms of tumor debulking is performed in order to promote survival

SUMMARY:
Extensive tumour debulking challenges both surgeon and anaesthesiologist but promotes survival in late-stage ovarian cancer patients. Little is known about the intraoperative fluid balance and its impact on morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for cytoreductive surgery in ovarian cancer

Exclusion Criteria:

* Age < 18 years
* unability to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
fluid balance | at the end of surgery
  intraoperative fluid balance is determined by the difference between fluid intake and outtake

SECONDARY OUTCOMES:
mechanical ventilation | at the timepoint of extubation
  Duration of mechanical ventilation, starting from endotracheal intubation until extubation
mortality | 5 years
  long-term mortality after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Soehle, MD, PhD, Principal Investigator — University Clinic Bonn
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No